CLINICAL TRIAL: NCT01578486
Title: Salsalate as an Adjunctive Treatment for Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Xiaoduo Fan, Principal Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-P-000798
Record Dates: First submitted 2012-04-11; First posted 2012-04-17 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Cognition; Metabolism; Antipsychotics; Psychopathology
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — salicylsalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- salsalate (Experimental): open-label trial of salsalate 3g/day
  Interventions: Drug: salsalate

INTERVENTIONS:
Drug: salsalate — open-label trial of salsalate 3g/day for 12 weeks.

SUMMARY:
This is a 12-week, open-label trial of salsalate 3 g/day as an adjunctive treatment in 15 schizophrenia subjects to examine salsalate's effect on psychopathology, cognitive functioning, and metabolic parameters.

Potential subjects will be identified by their clinicians at the Freedom Trail Clinic, or Massachusetts General Hospital. A total of 15 subjects will be enrolled.

DETAILED DESCRIPTION:
The specific aims include:

Primary aims:

1. Examine the efficacy of salsalate (3g/day) in improving positive and negative symptoms as measured by the Positive and Negative Syndrome Scale (PANSS) and the Scale for Assessment of Negative Symptoms (SANS).
2. Examine the efficacy of salsalate in improving cognition as measured by the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) composite score.

Secondary aims:

1. Examine salsalate's effects on inflammatory markers such as high sensitivity C-reactive protein (hs-CRP), TNF-α and IL-6.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Diagnosis of schizophrenia or schizoaffective disorder;
* Stable dose of the current antipsychotic drug for at least one month;
* Well established compliance with outpatient treatment per treating clinician's judgment;
* Able to complete the cognitive assessment battery (must be English speaking);
* Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods during the study.

Exclusion Criteria:

* Inability to provide informed consent;
* Current substance abuse;
* Psychiatrically unstable per treating clinician's judgment;
* Significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases;
* Currently on immunosuppressant medication including oral steroids;
* Use of anti-coagulants (heparin, LMWH, warfarin, cilostazol, clopidogrel, dabigatran);
* History of chronic infection (including, HIV and hepatitis), malignancy, organ transplantation, blood dyscrasia, central nervous system demyelinating disorder, and any other known autoimmune or inflammatory condition;
* Experienced asthma, urticaria or allergic type reaction after taking aspirin, salsalate, or other NSAIDS;
* Pregnancy or breastfeeding;
* Pre-existing chronic tinnitus.
* Known hypersensitivity to salsalate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, MPH, MS, Principal Investigator — UMass Medical School; Matthew R Goodnow, BS, Study Director — UMass Medical School
Locations (1):
- University of Massaschusetts Medical School, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 17 subjects consented and were screened, 4 of which were screen fails. The remaining 13 received the study medication.
Period: Overall Study
Arm/Group | Salsalate
Started | 13
Completed | 8
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Salsalate
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: PANSS Total Score
Description: Positive and negative symptoms of schizophrenia will be measured by total score on all subscales of the Positive and Negative Syndrome Scale (PANSS; score range 30-210). Higher scores correspond with worse outcomes.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Salsalate
Number analyzed (Participants) | 8
units on a scale
  Baseline | 58.2 (11.4)
  Week 12 | 53.5 (11.9)

2. Primary Outcome: SANS Total Score
Description: Negative symptoms of schizophrenia will be measured by total score on the Scale for Assessment of Negative Symptoms (SANS; score range 0-100). Higher scores correspond with worse outcomes.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Salsalate
Number analyzed (Participants) | 8
units on a scale
  Baseline | 33.0 (15.7)
  Week 12 | 33.0 (12.9)

3. Primary Outcome: MATRICS Composite Score
Description: Improved cognition will be measured using the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) assessment. The MATRICS assessment includes a battery of tests, and the composite t-score measures cognition across 7 domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. A higher score indicates better cognition.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Salsalate
Number analyzed (Participants) | 8
t-score
  Baseline | 27.9 (11.9)
  Week 12 | 31.6 (15.2)

4. Primary Outcome: PANSS Positive Score
Description: Subscale of Positive and Negative Syndrome Scale that specifically measures positive symptoms. The scores range from 7-49, with higher scores representing a worse outcome.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Salsalate
Number analyzed (Participants) | 8
units on a scale
  Baseline | 13.0 (5.4)
  Week 12 | 10.9 (4.4)

5. Primary Outcome: PANSS- Negative Score
Description: Subscale of Positive and Negative Syndrome Scale that specifically measures negative symptoms. The scores range from 7-49, with higher scores representing a worse outcome.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Salsalate
Number analyzed (Participants) | 8
units on a scale
  Baseline | 18.5 (6.5)
  Week 12 | 17.4 (6.1)

6. Secondary Outcome: Hs-CRP
Description: High-sensitivity C-reactive protein (hs-CRP) will be measured in mg/L in order to detect inflammation. Higher hs-CRP values correspond to higher levels of inflammation.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Salsalate
Number analyzed (Participants) | 8
mg/L
  Baseline | 3.0 (1.2)
  Week 12 | 2.0 (1.2)

7. Secondary Outcome: TNF-alpha
Description: Tumor necrosis-alpha factor will be measured to assess inflammation levels.
Time Frame: Baseline,12 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Salsalate
Number analyzed (Participants) | 8
pg/ml
  Baseline | 8.2 (3.7)
  Week 12 | 8.7 (3.6)

8. Secondary Outcome: IL-6
Description: IL-6 (interleukin 6) is a marker used to measure inflammation.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salsalate
Number analyzed (Participants) | 8
pg/mL
  Baseline | 2.2 (0.87)
  Week 12 | 2.3 (1.00)

ADVERSE EVENTS:
Arm/Group | Salsalate
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=8)
Stomach/Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Nausea/Vomiting (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Weakness (General disorders) | 1 (1)
Bloody urine (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No